CLINICAL TRIAL: NCT05413954
Title: To Evaluate the Health Effect of Particular Fatty Acids Profiles From Eggs
Acronym: Omegasnack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Omegasnack
Record Dates: First submitted 2022-05-30; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control snack
  Interventions: Other: Control
- Test (Experimental): Test snack
  Interventions: Other: Test

INTERVENTIONS:
Other: Control — Control group ate snacks composed of dried vegetables, one classical egg yolk and 2.3g of sunflower oil during 10 weeks
  Arms: Control
Other: Test — Tes group ate snacks composed of dried vegetables, one test egg yolk naturally enriched in rumenic acid, docosahexaenoic acid and punicic acid, 0.34g of pomegranate seed oil and 2.26g of olive oil during 10 weeks
  Arms: Test

SUMMARY:
In a previous study, 24 volunteers consumed two conventional eggs or two eggs naturally enriched with omega 3, 5 and 7 every day for 3 months. It was shown that these eggs were well tolerated and that the omega enrichment led to a reduction in waist circumference of 3 cm in 3 months.

The objective of Omegasnack study was therefore to go further in the evaluation of these effects on waist circumference; 1) confirm the effects of these eggs on waist circumference when included in a snack, 2) determine whether this reduction in waist circumference is linked to a reduction in muscle and/or fat mass (subcutaneous and/or visceral) and 3) evaluate whether these effects are associated with a modification in the accumulation of ectopic fat in the muscle and/or liver.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 75 years;
* Abdominal obesity: waist circumference for men > 94cm and > 80cm for women;
* Body mass index ≥ 25kg/m2 and ≤30kg/m2;
* For women: use of effective contraception;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* French speaker.

Exclusion Criteria:

* Uncontrolled systolic blood pressure > 160/100 mmHg;
* For premenopausal women: pregnant women or women planning to get pregnant within 3 months or lactating women;
* For menopausal women: less than 6 months of menopause;
* For Perimenopausal women: presenting symptoms;
* Type II diabetes (controlled or uncontrolled), Type I diabetes;
* Medical history or actual cardiovascular disease (myocardial infarction, angina, transient ischemic attack, lower limb arteriopathy);
* Medical history or actual severe psychiatric, hepatic, pancreatic, kidney, pulmonary or gastrointestinal problem
* Thyroid disorder;
* Cancer < 3 years before the screening visit;
* Smokers or who have stopped smoking within the last 6 months before the screening visit;
* Subject presenting allergy or food intolerance to eggs;
* Subjects who are not able to understand and follow study procedures;
* Drug addiction problem (regular consumption);
* Recent change of body weight > 7% (< 2 months before the inclusion);
* Within 1 month before the screening visit, change in the chronic (> 7 days in a row) intake or dosage of drug(s) or product(s) modifying the glucose and/or lipid metabolism;
* Current or recent (< 2 months before the screening visit) intake of dietary supplements rich in n-3 polyunsaturated fatty acid (including tablets, pills, capsules, enriched-oils);
* Vegan diet;
* Consumption of fish > 3 times per week;
* Women who drink more than 2 glasses of alcohol per day (> 20 g of alcohol per day or > 140g/week) or men who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day or more than 210g/week);
* LDL > 159 mg/dl or Total cholesterol > 239 mg/dl;
* Subjects having participated to another clinical trial < 1 month before the screening test visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of waist circumference at 10 weeks | Baseline, 10 weeks
Change from baseline of waist circumference at 5 weeks | Baseline, 5 weeks

SECONDARY OUTCOMES:
Satiety | Baseline, 5 weeks, 10 weeks
  Visual analog scale (between 0 = no satiety to 100 = complete satiety)
Red blood cells fatty acid pattern | Baseline, 5 weeks, 10 weeks
Plasma fatty acid pattern | Baseline, 5 weeks, 10 weeks
Plasma triglyceride | Baseline, 5 weeks, 10 weeks
Plasma LDL cholesterol | Baseline, 5 weeks, 10 weeks
Plasma total cholesterol | Baseline, 5 weeks, 10 weeks
Plasma HDL cholesterol | Baseline, 5 weeks, 10 weeks
Plasma non-HDL cholesterol | Baseline, 5 weeks, 10 weeks
Glycemia | Baseline, 5 weeks, 10 weeks
Insulinemia | Baseline, 5 weeks, 10 weeks
HOMA (Homeostatic Model Assessment for Insulin Resistance) | Baseline, 5 weeks, 10 weeks
QUICKI | Baseline, 5 weeks, 10 weeks
Body weight | Baseline, 5 weeks, 10 weeks
Impedancemeter lean mass | Baseline, 5 weeks, 10 weeks
Impedancemeter fat mass | Baseline, 5 weeks, 10 weeks
Hip circumference | Baseline, 5 weeks, 10 weeks
CRP (c-reactive protein) | Baseline,10 weeks
Oxidized LDL | Baseline,10 weeks
Endothelial status | Baseline,10 weeks
  HbNO (hemoglobin-NO adduct)
Liver stiffness | Baseline,10 weeks
  Transient elastography
Liver steatosis | Baseline,10 weeks
  Controlled attenuation parameter (CAP)
Subcutaneous fat area evaluated by computed tomography (CT) scan | Baseline,10 weeks
Visceral fat area evaluated by computed tomography (CT) scan | Baseline,10 weeks
Skeletal muscle index (total skeletal muscle area normalized for stature) evaluated by computed tomography (CT) scan | Baseline,10 weeks
Muscular radiation attenuation (fat accumulation in muscle) evaluated by computed tomography (CT) scan | Baseline,10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain - CICN, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No